CLINICAL TRIAL: NCT04112043
Title: Nicotinamide Riboside as an Enhancer of Exercise Therapy in Hypertensive Older Adults (The NEET Trial)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB201900746 -N-R; OCR26682 (Other: UF OnCore); 5R21AG064282 (NIH); AWD06755 (Other: UFIRST)
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Hypertension
Keywords: systolic blood pressure (SBP); cardiovascular (CV) disease
MeSH Terms: conditions — Hypertension; Disease | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NR plus Walking Exercise (Active Comparator): 1,000 mg/day of NR combined with three days/week of supervised, center-based walking exercise (n=18)
  Interventions: Behavioral: Walking Exercise; Drug: Nicotinamide Riboside (NR)
- Walking Exercise plus Placebo (Active Comparator): 1,000 mg/day of Placebo combined with three days/week of supervised, center-based walking exercise (n=18)
  Interventions: Behavioral: Walking Exercise
- NR Alone (Active Comparator): 1,000 mg/day of NR
  Interventions: Drug: Nicotinamide Riboside (NR)

INTERVENTIONS:
Behavioral: Walking Exercise — Participants randomized to this intervention 3 days/week of supervised, center-based walking exercise.
  Arms: NR plus Walking Exercise; Walking Exercise plus Placebo
Drug: Nicotinamide Riboside (NR) — Participants randomized to this intervention will receive 1,000 mg/day of NR.
  Arms: NR Alone; NR plus Walking Exercise

SUMMARY:
More than 80% of older adults have hypertension, with higher prevalence of high systolic blood pressure (SBP) putting them at high risk for cardiovascular (CV) disease and death. Novel compound, nicotinamide riboside may enhance the effects of exercise therapy in hypertensive older adults.

DETAILED DESCRIPTION:
More than 80% of older adults have hypertension, with a higher prevalence of high systolic blood pressure (SBP) putting them at high risk for cardiovascular (CV) disease and death. Because drug therapy that lowers SBP is associated with side effects such as hypotension, syncope, and kidney dysfunction, there is a great need for effective lifestyle SBP-lowering interventions for the older population that can replace drug therapy. While aerobic exercise is a recommended lifestyle intervention for controlling SBP and preventing CV disease naturally, in older adults it has been shown to be less effective in vascular-tissue remodeling because of arterial stiffness, resulting in less efficient SBP control. Reduced bioavailability of nicotinamide adenine dinucleotide (NAD+), a cofactor for the deacetylase sirtuin1 (SIRT1), may contribute to age-related vascular dysfunction via oxidative stress and reduced nitric oxide (NO). Exercise-induced overexpression of NAD+-dependent SIRT1 improves the bioavailability of NO. Preclinical evidence suggests that poor vascular function improvement in response to exercise in older mice is caused by insufficient NAD+ levels to stimulate SIRT1 activity. Importantly, replenishment of NAD+ levels induced vascular remodeling, improved vascular function, and reduced SBP in mice. An objective of this study, therefore, is to test a combination of aerobic exercise and nicotinamide riboside, a compound that replenishes NAD+ levels, to optimize exercise's SBP-lowering effect in hypertensive older adults. Initial human clinical trials demonstrated that nicotinamide riboside supplementation (1,000 mg/day) was safe and showed a higher potential to reduce SBP and arterial stiffness in participants with elevated SBP. As we have preclinical evidence that combining NAD+ replenishment with exercise is an ideal strategy for improving vascular function, our central hypothesis is that the intervention of aerobic-exercise training combined with nicotinamide riboside supplementation will reduce SBP in hypertensive older adults more effectively than will exercise alone. We will enroll 54 participants ≥ 55 years and older into either: (1) 1,000 mg/day of nicotinamide riboside plus 3 days/week of supervised, center-based walking exercise (n=18), or (2) the same exercise program combined with placebo (n=18), or (3) 1,000 mg/day of nicotinamide riboside alone (n=18). All participants will undergo daytime continuous SBP at baseline, 3 weeks, and 6 weeks, and arterial-stiffness measurements by pulse-wave velocity at baseline and at 6 weeks. Elevated SBP will be determined as daytime average equal to or above 130 mmHg, measured by the 24-hour blood-pressure device. To our knowledge, this study will be the first attempt to enhance exercise therapy with nicotinamide riboside in hypertensive older adults. We believe that nicotinamide riboside is "the missing piece of the puzzle" in improving vascular remodeling and SBP management in older adults. Preliminary evidence from this pilot study may support a full-scale Phase III clinical trial in hypertensive older adults. The ultimate goal of this line of research is to find adjuvant strategies to improve the exercise's SBP-lowering effects in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years and older
* Daytime average of systolic blood pressure of ≥ 130 mmHg and < 160 mmHg.
* Sedentary lifestyle, defined as < 150 min/wk of moderate physical activity as assessed by the CHAMPS questionnaire.
* Willingness to be randomized to either treatment group
* Willingness to participate in all study procedures

Exclusion Criteria:

* Failure to provide informed consent.
* Pregnant
* Change in blood pressure therapy (type or dose) within the last 3 months- Temporary Exclusion
* Daytime average of systolic blood pressure ≥160 mmHg.
* Regular consumption of nicotinamide riboside supplement
* Current involvement in supervised rehabilitation program
* Absolute contraindication(s) to exercise training according to American College of Sports Medicine guidelines [11]
* Daytime average of systolic blood pressure below 130mm Hg or Diastolic BP ≥ 100mm Hg.
* Peripheral vascular disease; peripheral neuropathy; retinopathy
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina;
* Myocardial infarction or stroke within past year
* Significant cognitive impairment, including known dementia diagnosis or a Mini-Mental State Examination exam score < 24
* Progressive, degenerative neurologic disease, e.g., Parkinson's Disease, multiple sclerosis;
* Severe rheumatologic or orthopedic diseases, e.g., awaiting joint replacement, active inflammatory disease;
* Severe pulmonary disease, requiring steroid therapy or the use of supplemental oxygen;
* Hip fracture, hip or knee replacement, or spinal surgery within past 4 months;
* Other significant co-morbid conditions that would impair ability to participate in the exercise-based intervention
* Simultaneous participation in another intervention trial

Ages: 55 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Mankowski, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Institute on Aging, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 147 enrolled participants, 54 met the eligible criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | NR Plus Walking Exercise | Walking Exercise Plus Placebo | NR Alone
Started | 17 | 18 | 19
Completed | 15 | 16 | 18
Not Completed | 2 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Taking NR supplement | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NR Plus Walking Exercise | Walking Exercise Plus Placebo | NR Alone | Total
Number analyzed (Participants) | 17 | 18 | 19 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (7.0) | 68.3 (7.7) | 66.3 (7.2) | 67.3 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 12 | 33
  Male | 6 | 8 | 7 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 6 | 15
  White | 12 | 13 | 11 | 36
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 18 | 19 | 54
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 33.0 (7.2) | 30.8 (5.7) | 30.7 (7.8) | 31.5 (6.9)
Baseline average daytime systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure was measured every 20 minutes (min) during the day (from 0700 to 2200 hours) at the baseline visit. Average daytime systolic blood pressure was calculated based on all the available daytime blood pressure readings recorded by the ambulatory blood pressure monitor. Population: Average daytime systolic blood pressure was calculated based on all the available daytime blood pressure readings recorded by the 24-hour ambulatory blood pressure monitor.
  mmHg | 138.5 (11.8) | 141 (12.1) | 138.8 (14.9) | 139.4 (12.8)
Baseline average daytime diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure was measured every 20 minutes (min) during the day (from 0700 to 2200 hours) at the baseline visit. Average daytime diastolic blood pressure was calculated based on all the available daytime blood pressure readings recorded by the ambulatory blood pressure monitor. Population: Average daytime diastolic blood pressure was calculated based on all the available daytime blood pressure readings recorded by the 24-hour ambulatory blood pressure monitor.
  mmHg | 75.5 (8.6) | 75.2 (6.5) | 78.2 (10.2) | 76.3 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Daytime Systolic Blood Pressure
Description: The primary outcome of this study is the change in average daytime systolic blood pressure. Systolic blood pressure was measured every 20 minutes (min) during the day (from 0700 to 2200 hours) at baseline and week 6 visits. Based on the American Heart Association guideline, we selected twenty valid daytime blood pressure recordings to calculate the average daytime value, then we calculated the mean differences between week 6 and baseline.
Time Frame: Baseline; Week 6
Population: Considering within-group differences for interested variables; we focus on the mean differences between week 6 and the baseline.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | NR Plus Walking Exercise | Walking Exercise Plus Placebo | NR Alone
Number analyzed (Participants) | 15 | 16 | 17
mmHg | 5.19 [-2.16 to 12.54] | -2.71 [-8.29 to 2.87] | -0.48 [-4.85 to 3.89]

2. Secondary Outcome: Change in Arterial Stiffness
Description: The measurement of aortic pulse-wave velocity (PWV), particularly between the carotid and femoral arteries (cfPWV), was conducted using the SphygmoCor XCEL system. Briefly, cfPWV was determined by recording pressure pulse waves at the carotid and femoral arteries using a high-fidelity micromanometer and calculating the distance between the recording sites divided by the time delay between the carotid and the femoral pulse waves.
Time Frame: Baseline; Week 6
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: m/s
Arm/Group | NR Plus Walking Exercise | Walking Exercise Plus Placebo | NR Alone
Number analyzed (Participants) | 14 | 15 | 16
m/s | -0.29 [-0.74 to 0.17] | -0.15 [-0.59 to 0.29] | -0.10 [-0.56 to 0.37]

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: We collected adverse events at baseline, 3-week visits, 6-week visits, and every exercise session.
Arm/Group | NR Plus Walking Exercise | Walking Exercise Plus Placebo | NR Alone
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18 | 1/19
Other Adverse Events (participants affected / at risk) | 9/17 | 12/18 | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NR Plus Walking Exercise (N=17) | Walking Exercise Plus Placebo (N=18) | NR Alone (N=19)
Sepsis and Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NR Plus Walking Exercise (N=17) | Walking Exercise Plus Placebo (N=18) | NR Alone (N=19)
Pancytopenia Worsening (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Felt "spasm" feeling in the stomach (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headaches, loose stool, dry mouth and nose, fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
High blood sugar (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
High PSA , high creatinine, frequent urination, increased hunger (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sciatic Nerve Pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Knee Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Hurt Foot/Leg at Home (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Soreness from Exercise (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Symptoms (difficulty breathing, headache, etc.) due to COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Allergies Became Worse (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tripped and fell (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Cold or flu with symptoms (sneezing, runny nose, congestion, etc.) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Irregular Heartbeat (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Change in diabetes symptoms (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
UTI (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cyst removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bloody Urine (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus problems (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Annoying feeling at the bottom of both feet due to calluses (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT04112043/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT04112043/ICF_001.pdf